CLINICAL TRIAL: NCT02633644
Title: The Harmony System for the Treatment of Heart Failure Patients - A Safety and Performance Study
Brief Title: Endovascular NeuromoDulation Treatment fOr Heart Failure Patients (ENDO-HF)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The company shut down
Sponsor: Enopace Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-250
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure
Keywords: Heart Failure; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treated with Harmony System (Experimental): Implantation and activation of the Harmony endovascular neurostimulator
  Interventions: Device: Harmony System

INTERVENTIONS:
Device: Harmony System — Percutaneous neuromodulation of the aortic wall

SUMMARY:
The purpose of the ENDO-HF study is to determine the safety & performance of the Harmony System for the treatment of heart failure

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed as chronic heart failure NYHA class II-III
* Subject should be receiving optimal medical treatment
* Subject signed and dated informed consent

Exclusion Criteria:

* Subject has severe aortic sclerosis or calcification
* Subject diagnosed with severe aortic valve disease
* Subject has severe mitral stenosis
* Subject involved in any concurrent clinical investigation
* Subject with cerebral vascular accident or transient ischemic attack prior to enrollment
* Subject diagnosed with Marfan Syndrome
* Subject with moderate or severe chronic obstructive lung disease
* Subject is allergic to iodine or contrast media
* Subject with prior cardiac transplant or heart transplant candidate
* Subject with a life expectancy of less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
The occurrence of all system and/or procedure related serious adverse events | 6 months

SECONDARY OUTCOMES:
The change in the New York Heart Association (NYHA) functional class as set by the Primary Investigator (PI) | 6 months
The change in the exercise capacity as defined in a 6-minute walk test | 6 months
The change in heart failure symptoms, as measured by quality of life, defined as an improvement from baseline on the Minnesota Living with Heart Failure® Questionnaire (MLWHFQ) | 6 months
The change in echocardiographic assessment of LV ejection fraction | 6 months
The change in echocardiographic assessment of LV end systolic volume | 6 months
The change in echocardiographic assessment of LV end diastolic volume | 6 months
The change in echocardiographic assessment of left atrium volume index | 6 months
The change in echocardiographic assessment of LV mass index | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weiss, MD, Study Director — Enopace Biomedical
Locations (5):
- OLV Hospital, Aalst, Belgium
- University Hospital Center Zagreb, Zagreb, Croatia
- Hippokration General Hospital, Athens, Greece
- Israel (2):
  - Rambam Healthcare Campus, Haifa
  - Baruch Padeh Medical Center (Poriya), Tiberias